CLINICAL TRIAL: NCT06659926
Title: 68Ga-PSMA-PET/CT and Genomic Alterations for Future Selection of Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC) for Radium-223 Treatment.
Brief Title: The Radium-select Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M24PSM; NL86928.041.24 (Registry Identifier: ABR formulier)
Record Dates: First submitted 2024-08-16; First posted 2024-10-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: mCRPC; Male Urogenital Diseases
Keywords: mCRPC; 68Ga-PSMA-PET/CT; Radium-223; Bone only-disease
MeSH Terms: conditions — Male Urogenital Diseases | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a prospective clinical study in which patients with mCRPC and bone-only disease according to ceCT and bone scan will receive standard-of-care treatment with Radium-223. In addition to standard-of-care systemic treatment, each patient will undergo an additional 68Ga-PSMA-PET/CT scan at baseline and will be followed throughout the treatment with online patient reported outcome measure (PROM) questionnaires (Kaiku application) and blood sampling for circulating tumor DNA (ctDNA) analysis.
Masking Description: The treating physicians will be blinded to the result of the baseline 68Ga-PSMA-PET/CT scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mCRPC patients with bone-only disease according to 68Ga-PSMA-PET/CT (Other): a prospective clinical study in which patients with mCRPC and bone-only disease according to ceCT and bone scan will receive standard-of-care treatment with Radium-223. In addition to standard-of-care systemic treatment, each patient will undergo an additional 68Ga-PSMA-PET/CT scan at baseline and will be followed throughout the treatment with online patient reported outcome measure (PROM) questionnaires (Kaiku application) and blood sampling for circulating tumor DNA (ctDNA) analysis.
  Interventions: Other: 68Ga-PSMA-PET/CT scan

INTERVENTIONS:
Other: 68Ga-PSMA-PET/CT scan — 68Ga-PSMA-PET/CT scan at baseline and will be followed throughout the treatment with online patient reported outcome measure (PROM) questionnaires (Kaiku application) and blood sampling for circulating tumor DNA (ctDNA) analysis. At clinical progression, each patient will undergo a second 68Ga-PSMA-PET/CT to determine the location of disease progression and assess the value of 68Ga-PSMA-PET/CT imaging as a response measure
  Other Names: Online patient reported outcome measure (PROM) questionnaires; Blood sampling

SUMMARY:
Radium-223 is an established radionuclide therapy for patients with metastatic castration resistant prostate cancer (mCRPC) and symptomatic bone metastasis. Patients are eligible for this treatment when they have mCRPC and bone metastases; limited extraskeletal lesions (local prostate, lymph nodes <3 cm) on conventional contrast enhanced CT (ceCT) were allowed in the registration trial(1). Previous research revealed that extraskeletal disease on ceCT and bone scans correlates with a poor response. Meanwhile, 68Ga-PSMA-PET/CT emerged as more sensitive imaging strategy that increases the detection of extraskeletal prostate cancer metastases. It is unclear whether these extraskeletal lesions harbour any predictive value in the treatment of mCRPC patients with Radium-223.

DETAILED DESCRIPTION:
Study design:

The investigators will conduct a prospective clinical study in which patients with mCRPC and bone-only disease according to ceCT and bone scan will receive standard-of-care treatment with Radium-223. In addition to standard-of-care systemic treatment, each patient will undergo an additional 68Ga-PSMA-PET/CT scan at baseline and will be followed throughout the treatment with patient reported outcome measure (PROM) questionnaires (Kaiku application) and blood sampling for circulating tumor DNA (ctDNA) analysis. The treating physicians will be blinded to the result of the baseline 68Ga-PSMA-PET/CT scan. Each patient will receive a maximum number of 6 cycles of Radium-223 therapy according to current clinical guidelines and will undergo response evaluation by ceCT and bone scans upon clinical progression. At clinical progression, each patient will undergo a second 68Ga-PSMA-PET/CT to determine the location of disease progression and assess the value of 68Ga-PSMA-PET/CT imaging as a response measure. The clinical response of Radium-223 therapy in the patients with bone-only disease according to 68Ga-PSMA-PET/CT scanning, will be compared to the treatment outcomes collected in our previously reported ROTOR registry. Secondary aims are to determine the value of ctDNA as predictive biomarker and the value of 68Ga-PSMA-PET/CT imaging in the response assessment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Progressive disease after previous treatment defined as a rise in serum (Prostate Specific Antigen) PSA (PCWG3 criteria(22), see appendix 1) and/or progression on conventional imaging (PCWG3).
* A positive bone scan (osteoblastic bone metastases), with at least two metastases.
* Hemoglobin concentration >10 g/dl (6.2 mmol/l) and thrombocytes >100 109/I at baseline.
* Each patient will need to (continue to) receive adequate bone protective agents (e.g. bisphosphonates) and androgen deprivation therapy (ADT) according to current clinical guidelines.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance score >2
* Life expectancy < 6 months.
* Detected extra-skeletal metastases or lymph node metastases (>3 cm short axis) as identified by conventional imaging (ceCT thorax/abdomen)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical progression free survival (cPFS) | Up to 28 weeks
  The primary study endpoint will be clinical progression free survival (cPFS) in 30 patients with bone-only disease according to PSMA PET/CT.

SECONDARY OUTCOMES:
Patient reported outcome measures ( PROMs). | In screening and cycle 2,3,4,5,6 (every 4 weeks) and with progression
  complete questionnaires on health related quality of life (HRQoL), including the (Functional Assessment of Cancer Therapy) FACT-P: Score 1 to 4, Brief pain Inventory (BPI-SF): scale score from 1 to 10, and analgesics use; name, dosing, frequence and after every treatment cycle.
Overall survival (OS) | In Follow up (q6months, max 24 months)
  OS will be defined as time from first Radium-223 treatment to the date of death, or censored at last follow-up.
Baseline and changes in 68 Ga-PSMA-PET-CT parameters | Baseline and until progression
  Baseline and changes in 68Ga-PSMA-PET/CT parameters (disease localizations, extent of disease, tumor volume).
Genomic biomarkers in ctDNA | Before treatment, cycle 3 and 5 and with progression
  We will determine whether homologous recombination deficiency (HRD) assessment in ctDNA correlates with a favorable therapy response. We will perform deep whole genome sequencing (WGS) of ctDNA to determine the clonal evolution of prostate cancer during Radium-223 therapy.

CONTACTS AND LOCATIONS:
Overall Officials: J.C. van der Mijn, Principal Investigator — NKI-AvL
Locations (5):
- Netherlands (5):
  - NKI-AVL, Amsterdam, North Holland
  - Meander Medisch Centrum, Amersfoort, Utrecht
  - Sint Antonius ziekenhuis, Nieuwegein, Utrecht
  - Diakonessenhuis, Utrecht
  - UMC, Utrecht

IPD SHARING:
Plan to Share IPD: No